CLINICAL TRIAL: NCT02188550
Title: Phase II Single Arm Trial With Combination of Everolimus and Letrozole in Treatment of Platinum Resistant Relapse or Refractory or Persistent Ovarian Cancer/Endometrial Cancer (CRAD001CUS242T)
Brief Title: Single Arm Trial With Combination of Everolimus and Letrozole in Treatment of Platinum Resistant Relapse or Refractory or Persistent Ovarian Cancer/Endometrial Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sinai Hospital of Baltimore (Other)
Responsible Party: Principal Investigator, Kenneth Miller, M.D., Medical Oncologist, Sinai Hospital of Baltimore
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001CUS242T
Record Dates: First submitted 2014-05-09; First posted 2014-07-11 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Ovarian Cancer; Endometrial Cancer
Keywords: relapse or refractory or persistent epithelial ovarian fallopian tube; primary peritoneal carcinoma or endometrial cancer
MeSH Terms: conditions — Ovarian Neoplasms; Endometrial Neoplasms; Recurrence | interventions — Everolimus; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single (Experimental): This is a single arm, non-randomized, open-label study with a combination of everolimus and letrozole once a day dosing . Each cycle would be 28days and patients would be scanned after every 3 cycles for response, until disease progression is documented
  Interventions: Drug: everolimus and letrozole

INTERVENTIONS:
Drug: everolimus and letrozole — This is a single arm, non-randomized, open-label study with a combination of everolimus and letrozole once a day dosing . Each cycle would be 28days and patients would be scanned after every 3 cycles for response, until disease progression is documented
  The duration of the study will be until disease progression
  Everolimus and Letrozole will be administered as noted below;
  6.1.1 Dosing regimen
  Dosage : Everolimus Dose: 10 Unit: mg Frequency: daily Route of administration: Orally Dosage : Letrozole Dose: 2.5 Unit: mg Frequency: daily Route of administration: Orally

SUMMARY:
The purpose of the study is to determine if the combination of Everolimus and Letrozole is effective in the treatment of women with either recurrent or persistent epithelial ovarian, fallopian tube, primary peritoneal or endometrial cancer.

Experiments have shown that everolimus (Afinitor®) can prevent cells such as cancer from growing in number. Therefore, everolimus (Afinitor®) is being tested in specific diseases to stop cells from growing too fast (as in cancer).

Everolimus (Afinitor®) has been FDA approved for adults with advanced kidney cancer (Renal Cell Carcinoma). Everolimus (Afinitor®) received approval for patients with subependymal giant cell astrocytoma (SEGA), a brain tumor seen with genetic conditions called tuberous sclerosis complex (TSC) who require therapy, but are not candidates for surgery. Everolimus (Afinitor®) was approved for pancreatic neuroendocrine tumor (PNET) in patients with unresectable, locally advanced, or metastatic disease. Everolimus (Afinitor®) received approval for the treatment of postmenopausal women with advanced hormone receptor-positive, HER2- negative breast cancer (advanced HR+ BC) in combination with exemestane, after failure of treatment with letrozole or anastrozole. Everolimus (Afinitor®) also received approval for the treatment of patients with TSC who have renal angiomyolipoma not requiring immediate surgery.

Everolimus (Afinitor®) has been used to treat patients in clinical studies since 2002 and approximately 25,645 patients (as of 30-Sep-2012) have been treated with everolimus (Afinitor®).

DETAILED DESCRIPTION:
This is a single arm, non-randomized, open-label study with a combination of everolimus and letrozole once a day dosing . Each cycle would be 28days and patients would be scanned after every 3 cycles for response, until disease progression is documented.

Subjects will take two pills once a day by mouth with a glass of water.

Before the study…

Subjects will need to have the following exams, tests or procedures to find out if they can be in the study. These exams, tests or procedures are part of regular cancer care and may be done even if subjects do not join the study. If subjects have had some of them recently, they may not need to be repeated. This will be up to your study doctor.

* Medical history risk and physical examination,
* Blood tests to measure blood counts, blood mineral levels, and check liver and kidney function,
* CT scan or MRI of the abdomen and pelvis to measure detectable tumor
* A pregnancy blood test if subjects are capable of becoming pregnant
* Urinalysis (examination of urine)
* The European Organization for research and treatment of cancer global quality of life questionnaire C30 (QLQ-C30) -This standard questionnaire helps us to measure quality of life. This questionnaire will take subjects 15 minutes to complete and will be completed at entry into the study and at week 12 and 24 during the study.

Tests will be done for hepatitis B and/or C if:

* Subjects have a risk of having hepatitis B and/or C or if subjects live or have lived in specific geographical areas, such as Asia, Africa, Central and South America, Eastern Europe and Spain, Portugal or Greece;
* The study doctor thinks it is appropriate.

Subjects that have positive hepatitis B or hepatitis C results at screening may be required to take medication for up to 2 weeks before they start everolimus (Afinitor®) treatment.

During the Study…

If the exams, tests and procedures show that subjects can be in the study, and they choose to take part, then they will need the following tests and procedures. They are part of regular cancer care.

* History and physical examination
* Weekly blood tests to measure blood counts, blood mineral levels, blood clotting and check liver and kidney function
* Evaluation of side effects subjects may experience from the study treatment
* Tests to having hepatitis B and/or C
* CT scan or MRI of the abdomen and pelvis every 12 weeks
* The European Organization for research and treatment of cancer global quality of life questionnaire C30 (QLQ-C30)

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal or post-oophorectomy.
* Performance status Less than or equal to ECOG 2
* Patients must have relapse or refractory or persistent epithelial ovarian, fallopian tube, primary peritoneal carcinoma or endometrial cancer. Histologic documentation of the original primary tumor is required via pathology report.
* Patients must have received treatment with a platinum-based chemotherapeutic regimen for management of primary disease containing carboplatin, cisplatin. This initial treatment may have included intraperitoneal therapy, consolidation, noncytotoxic agents (biologic/targeted therapy) or extended therapy administered after surgical or non-surgical assessment.
* Patients must have platinum-resistant disease, defined as progression < 12 months after completion of first-or-second-line platinum based chemotherapy. The date (platinum-free interval) should be calculated from the last administered dose of platinum therapy.
* Platinum sensitive patients must have progressed/relapsed after receiving a second line platinum therapy.
* Patients with platinum-refractory primary disease, defined as having disease3 progression while receiving first-line platinum-based chemotherapy.
* Patients are allowed to receive, but are not required to receive, one additional cytotoxic regimen for management of relapse or refractory or persistent disease.
* Patients are allowed to have received, but are not required to have received, biologic/targeted therapy (e.g., bevacizumab and/or PARP inhibitor) as part of their primary treatment regimen or for management of relapse or refractory or persistent disease.

Exclusion Criteria:

* Patients currently receiving anticancer therapies or who have received anticancer therapies within 4 weeks of the start of Everolimus (including chemotherapy, antibody based therapy, etc.); radiation therapy within 2 weeks.
* Known intolerance or hypersensitivity to Everolimus or other rapamycin analogs (e.g.

sirolimus, temsirolimus) or to Letrozole.

* Known impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral Everolimus;
* Patients who have any severe and/or uncontrolled medical conditions such as:

  1. unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction ≤6 months prior to start of Everolimus, serious uncontrolled cardiac arrhythmia, or any other clinically significant cardiac disease
  2. Symptomatic congestive heart failure of New York heart Association Class III or IV
  3. active (acute or chronic) or uncontrolled severe infection, liver disease such as cirrhosis, decompensated liver disease, and active or chronic hepatitis (i.e. quantifiable HBV-DNA and/or positive HbsAg, quantifiable HCV-RNA),
  4. known severely impaired lung function (spirometry and DLCO 50% or less of normal and O2 saturation 88% or less at rest on room air),
  5. active, bleeding diathesis;
* Chronic treatment with corticosteroids or other immunosuppressive agents. Topical or inhaled corticosteroids are allowed;

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-06; Primary Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Tumor Response to treatment with Everolimus and Letrozole using RECIST Criteria | Baseline, Then every 12 weeks while on Everolimus and Letrozole up to 36 months
  The duration of response will be documented and also compared to the duration of response ot the last, most recent, cancer treatment.

SECONDARY OUTCOMES:
Overall survival of patients treated with the combination of letrozole and everolimus | From randomization until date of death, assessed up to 36 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sinai Hospital of Baltimore, Inc., Baltimore, Maryland, United States